CLINICAL TRIAL: NCT01688908
Title: Effcacy of Endoscopic Screening for Esophageal Cancer in China (ESECC): a Population-based Randomized Controlled Trial
Brief Title: Efficacy of Endoscopy Screening on Esophageal Cancer in China (ESECC)
Acronym: ESECC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Yang Ke, Professor, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 201202014
Record Dates: First submitted 2012-09-17; First posted 2012-09-20 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Esophageal Squamous Cell Carcinoma; Dysplasia
Keywords: Esophageal Squamous Cell Carcinoma; Endoscopic Screening; Efficacy; Cost-utility; High risk region; China
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Arm (No Intervention): Participants in this arm will not accept the endoscopic screening and only baseline and follow-up interview will be conducted in this arm.
- Screening Arm (Experimental): Participants in this arm will accept a baseline endoscopic screening, questionnaire investigation and follow-up interview. Subsequent re-examination and further medical services would be arranged among individuals who already have high-grade lesions found at baseline screening.
  Interventions: Procedure: Endoscopic Screening

INTERVENTIONS:
Procedure: Endoscopic Screening — 1. Upper G.I. endoscopic examination with Lugols Iodine in esophagus
  2. Biopsy at the visually abnormal sites
  3. Pathologic examination of all biopsy tissue specimens
  4. Subsequent re-examination and further medical services among individuals who already have high-grade lesions found at screening.
  5. Advises of endoscopic or surgical treatment will be given to participants who are diagnosed of high grade upper G.I. lesions.
  Arms: Screening Arm

SUMMARY:
To evaluate the efficacy of endoscopic screening on esophageal cancer (EC) and determine the most cost-effective strategy of endoscopic screening in high risk population in China, 668 villages of Hua county, a high risk area of esophageal cancer, were randomized into screening arm and control arm in a ratio of 1:1 and the total sample size is over 32,000 (~16,000 per group). Participants in the screening arm will accept standard chromoendoscopy examination to detect early esophageal cancer and no screening were designed in the control arm. The incidence of advanced EC, EC-specific mortality and all-cause mortality will be compared within the two groups to test the hypothesis that endoscopic screening would alter the natural history of lesions in esophagus and the incidence of advanced stage EC, EC-specific mortality and all-cause mortality in the screening arm will be lower than the control group. Cost-effectiveness analysis will also be conducted to find the most cost-effective strategy of endoscopic screening in rural China.

DETAILED DESCRIPTION:
BACKGROUND Esophageal cancer (EC) is one of the most common cancers in the world, and is a leading cause of cancer death, with more than 450,000 new cases and 400,000 deaths in 2012.Nearly half of the new cases of EC worldwide are found in China, and esophageal squamous cell carcinoma (ESCC) is the predominant histologic type. A series of etiologic factors for ESCC have been proposed in previous studies conducted in high prevalence regions of China, including age, family history of ESCC, poor nutritional status, smoking and drinking, chemical carcinogen exposure, and human papillomavirus (HPV) infection. But the main etiologic factors have not been definitively identified.

Because there are typically no symptoms in the early stages of ESCC, the vast majority of cases are clinically diagnosed at an advanced stage. The overall five-year survival is about 20% in China, and is even lower in less developed countries. However, if the disease is found at an early stage, the five-year survival may be 80% or greater. This profound improvement in survival indicates there is clearly a need for effective early detection strategies to enable earlier diagnosis and curative treatment. Esophageal squamous dysplasia (ESD) is considered to be the premalignant precursor lesion for ESCC, and harbors a high risk for progression into invasive cancer. ESD as well as early-stage malignant lesions (carcinoma in situ, CIS) are therefore screening targets for ESCC. Various screening methods have been tested, and endoscopy with iodine staining is the gold standard technique for the diagnosis of ESCC and its precursor lesions. Endoscopic screening has therefore been widely accepted as an optimal strategy in the secondary prevention of ESCC. However, taking the high cost and invasive nature of endoscopy into consideration, the efficacy and cost-effectiveness of such screening, must be evaluated prior to introduction of a population-wide screening program. Evidence regarding the efficacy of endoscopic screening for ESCC has been based predominantly on observational studies in high risk regions. There has been only one non-randomized controlled trial which reported that endoscopy plays a positive role in reducing mortality. No randomized controlled trials (RCTs) evaluating endoscopic screening have been reported to date. Observational studies and trials which are not randomized are limited in determining the true benefits of screening on reducing mortality due to potential lead-time bias, length-time bias and confounding bias. Hence, one-step large-scale population-based RCT are needed to determine the efficacy of endoscopic screening for ESCC.

In January 2012, we initiated the ESECC (Endoscopic Screening for Esophageal Cancer in China) trial in rural Hua County of Henan Province, which is a high-risk region in northern central China. This is the first population-based RCT aiming to evaluate the efficacy and cost-effectiveness of endoscopic screening for ESCC worldwide.

STUDY DESIGN Setting and participants This ESECC trial was undertaken in rural Hua County, which is an agricultural region in the northern part of Henan Province, Peoples Republic of China with a rural population of 1.1 million. The mortality for ESCC in this area is among the highest in the world.

Participants were eligible for the study if they meet the following criteria: 1) permanent residency in a target village; 2) age 45-69 (>5 years of life expectancy), and no history of endoscopic examination within 5 years prior to the initial interview; 3) no history of cancer or mental disorder; 4) negative for hepatitis B virus (HBV), hepatitis C virus (HCV) and human immunodeficiency virus (HIV); 5) voluntary participation and agreement to complete all phases of the examination.

Randomization This ESECC trial was designed as a cluster RCT. There are a total of 968 villages in rural Hua County, and 668 target villages were randomly selected from the 846 villages with population sizes ranging from 500 to 3,000 in Hua County. These 668 target villages were randomly allocated into the screening arm of the study or the control arm at a ratio of 1:1 (334 villages in each arm), using a blocked randomization procedure based on the total population size of each village for balancing the sample sizes between the two study arms.

Sample size According to the New Rural Cooperative Medical Scheme (NCMS) registration system of Hua County, the combined incidence rate of advanced esophageal cancer and cancer of the gastric cardia in the targeted population (age 45-69) was estimated to be 184.07/100,000 in 2011. Calculation of required sample size was based on the following assumptions: the average period of progression from severe dysplasia to EC is 5 years, and the accrual time is 5 years; the study period was set at 10 years, and 5% of the participants would be lost to follow-up per year; 5% of the participants in the control arm would seek endoscopic examination independently during the study period. Finally, with a total of 32,337 participants enrolled (1:1 between arms, ~20% of all eligible residents in target villages), statistical power of 86% at a one-sided 0.025 significance level can be achieved, even if only 30% of advanced EC cases were protected by screening. The number of participants enrolled in each target village was determined by the weight of the population size of the very village in the total population of the whole arm.

Intervention An informed consent was obtained from each study participant. Basic information including name, gender, date of birth, address and phone number was then collected and managed using a custom-designed database system. All participants received a physical examination which included measurement of height, weight and blood pressure. Blood samples were collected to screen for HBV, HCV and HIV, and participants with any of these infections were excluded. A computer aided one-on-one questionnaire investigation was conducted for all participants by trained interviewers to collect data on potential risk factors for esophageal cancer. EQ-5D-3L, a standardized generic instrument, was used in this ESECC trial to assess health related quality of life (HRQOL).Standardized explanations regarding the items in the questionnaire were provided if the participant was unable to understand the questions or respond appropriately.

In the screening arm, standard upper gastrointestinal endoscopy (UGE) with iodine staining was performed by physicians experienced in endoscopic examination. The entire esophagus and stomach were visually examined and biopsies were taken from all focal lesions. Standard sites in the esophagus (28 and 33 centimeters distal to the incisors in the 6 o'clock position) were biopsied if no visually identifiable abnormalities were found elsewhere. Biopsy specimens were fixed in 10% formaldehyde, embedded in paraffin, sectioned at 5μm, and stained with hematoxylin and eosin. The biopsy slides were reviewed by pathologists at Anyang Cancer Hospital without knowledge of the endoscopic findings. Diagnoses of ESD (mild, moderate and severe), CIS and squamous cell carcinoma were independently confirmed by two pathologists and discrepancies in their histologic diagnoses were adjudicated by consultation. To reflect the situation in real population-level screening as much as possible, participants who were diagnosed with severe squamous dysplasia, CIS or squamous cell carcinoma in the esophagus or malignant lesions in other sites were only informed of the diagnosis and provided with appropriate medical advice, rather than arranging directly for their further clinical treatment.

In the control arm, no endoscopic screening was performed and an abdominal ultrasound scan which had no association with the diagnosis of esophageal cancer was used.

Follow-up and outcomes The primary endpoint of the trial was EC-specific mortality, and the secondary endpoints included mortality from all causes, incidence of advanced EC and cost per quality-adjusted-life-year (QALY) gained. Two sources of follow-up data were used to identify outcome events in this study, namely door-to-door interviews, and electronic registry data. A record of vital events, including the experience of UGE, onset of cancer and death, will continue to be collected through annual door-to-door interviews with all cohort members. Data regarding cancer occurrence and death were also collected from the New Rural Cooperative Medical Scheme (NCMS) of Hua County, which is a government-run health insurance program in rural China with a nearly 100% participation rate which has been proved to be an ideal data source regarding cancer occurrence, diagnosis and treatment, and from the Death Registry of National Centers for Disease Control and Prevention (DR-CCDC) respectively.

Ethics statement This trial was approved by the Institutional Review Board of the Peking University School of Oncology, China. Informed consent was obtained from each participants.

ELIGIBILITY:
Participants were eligible for the study if they meet the following criteria: 1) permanent residency in a target village; 2) age 45-69 (>5 years of life expectancy), and no history of endoscopic examination within 5 years prior to the initial interview; 3) no history of cancer or mental disorder; 4) negative for hepatitis B virus (HBV), hepatitis C virus (HCV) and human immunodeficiency virus (HIV); 5) voluntary participation and agreement to complete all phases of the examination.

Ages: 45 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33948 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Esophageal cancer specific mortality | 5-10 years
Cost for saving 1 quality-adjusted life year (QALY) | 5-10 years

SECONDARY OUTCOMES:
Cumulative incidence of advanced esophageal cancer | 5-10 years
Change of life quality due to early diagnosis and treatment | 5-10 years

CONTACTS AND LOCATIONS:
Overall Officials: Yang Ke, M.D., Principal Investigator — Laboratory of genetics, Peking University cancer Hospital and institute
Locations (1):
- Laboratory of genetics, Peking University cancer Hospital and institute, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] He Z, Liu Z, Liu M, Guo C, Xu R, Li F, Liu A, Yang H, Shen L, Wu Q, Duan L, Li X, Zhang C, Pan Y, Cai H, Ke Y. Efficacy of endoscopic screening for esophageal cancer in China (ESECC): design and preliminary results of a population-based randomised controlled trial. Gut. 2019 Feb;68(2):198-206. doi: 10.1136/gutjnl-2017-315520. Epub 2018 Jan 6. PMID 29306867
- [Derived] He Z, Ke Y. Evolving diagnostic and surveillance strategies in esophageal cancer screening: Evidence from population-based studies in China. Chin J Cancer Res. 2025 Dec 30;37(6):929-936. doi: 10.21147/j.issn.1000-9604.2025.06.05. PMID 41523838
- [Derived] Wu M, Tian H, Guo C, Liu Z, Pan Y, Liu F, Liu Y, Yang W, Chen H, Hu Z, Liu M, He Z, Ke Y. Early-life undernutrition increases the risk of death from chronic diseases in adulthood: a population-based cohort study. Glob Health Res Policy. 2025 Jul 10;10(1):28. doi: 10.1186/s41256-025-00422-0. PMID 40635115
- [Derived] Liu M, Yang W, Guo C, Liu Z, Li F, Liu A, Yang H, Shen L, Wu Q, Duan L, Wang H, Tian H, Shi C, Pan Y, Liu Y, Liu F, Weiss NS, Cai H, He Z, Ke Y. Effectiveness of Endoscopic Screening on Esophageal Cancer Incidence and Mortality: A 9-Year Report of the Endoscopic Screening for Esophageal Cancer in China (ESECC) Randomized Trial. J Clin Oncol. 2024 May 10;42(14):1655-1664. doi: 10.1200/JCO.23.01284. Epub 2024 Mar 8. PMID 38457759
- [Derived] Zheng H, Liu Z, Chen Y, Ji P, Fang Z, He Y, Guo C, Xiao P, Wang C, Yin W, Li F, Chen X, Liu M, Pan Y, Liu F, Liu Y, He Z, Ke Y. Development and external validation of a quantitative diagnostic model for malignant gastric lesions in clinical opportunistic screening: A multicenter real-world study. Chin Med J (Engl). 2024 Oct 5;137(19):2343-2350. doi: 10.1097/CM9.0000000000002903. Epub 2024 Feb 26. PMID 38403900
- [Derived] Liu M, Qi Z, Zhou R, Guo C, Liu A, Yang H, Li F, Duan L, Shen L, Wu Q, Liu Z, Pan Y, Liu F, Liu Y, Cai H, He Z, Ke Y. How should extra-large Lugol-unstained lesions of the esophagus be treated? Results from a population-based cohort study. Cancer Med. 2023 Oct;12(19):20129-20139. doi: 10.1002/cam4.6592. Epub 2023 Sep 21. PMID 37732496
- [Derived] Liu Z, Liu M, Liu Y, Zhou R, Abliz A, Yuan W, Guo C, Zhang L, He W, Zheng H, Huang Y, Pan Y, Liu F, Hu Z, Chen H, Cai H, He Z, Ke Y. Absence of Lugol staining indicates initiation of esophageal squamous cell carcinoma: A combined genomic and epidemiologic study. Cell Rep Med. 2023 Sep 19;4(9):101168. doi: 10.1016/j.xcrm.2023.101168. Epub 2023 Aug 24. PMID 37625408
- [Derived] Hu N, Wang K, Zhang L, Liu ZJ, Jin Z, Cui RL, Zhang HJ, He ZH, Ke Y, Duan LP. Epidemiological and clinical features of functional dyspepsia in a region with a high incidence of esophageal cancer in China. Chin Med J (Engl). 2021 Jun 4;134(12):1422-1430. doi: 10.1097/CM9.0000000000001584. PMID 34091519
- [Derived] Wang MM, Guo CH, Li FL, Xu RP, Liu Z, Pan YQ, Liu FF, Liu Y, Cai H, Liu MF, He ZH, Ke Y. Family history of esophageal cancer modifies the association of serum lipids and malignant esophageal lesions: a nested case-control study from the "Endoscopic Screening for Esophageal Cancer in China" trial. Chin Med J (Engl). 2021 Apr 7;134(9):1079-1086. doi: 10.1097/CM9.0000000000001432. PMID 33840743
- [Derived] Li F, Li X, Guo C, Xu R, Li F, Pan Y, Liu M, Liu Z, Shi C, Wang H, Wang M, Tian H, Liu F, Liu Y, Li J, Cai H, Yang L, He Z, Ke Y. Estimation of Cost for Endoscopic Screening for Esophageal Cancer in a High-Risk Population in Rural China: Results from a Population-Level Randomized Controlled Trial. Pharmacoeconomics. 2019 Jun;37(6):819-827. doi: 10.1007/s40273-019-00766-9. PMID 30809788
- [Derived] Wang H, Pan Y, Guo C, Li F, Xu R, Liu M, Liu Z, Liu F, Cai H, Ke Y, He Z. Health-related quality of life among rural residents aged 45-69 years in Hua County, Henan Province, China: Results of ESECC Trial for esophageal cancer screening with endoscopy. Chin J Cancer Res. 2018 Apr;30(2):240-253. doi: 10.21147/j.issn.1000-9604.2018.02.07. PMID 29861609
- See also: Report of the design and preliminary results of the ESECC trial — https://www.ncbi.nlm.nih.gov/pubmed/29306867